CLINICAL TRIAL: NCT05144204
Title: Evaluation of Treatment Effect and Mechanism of Low FODMAP Diet in Treatment of Irritable Bowel Syndrome Patients
Brief Title: Evaluation of Treatment Effect of Low FODMAP Diet in Treatment of IBS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-07-023B
Record Dates: First submitted 2021-09-06; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: Low FODMAP diet
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irritable Bowel Syndrome Patients (Experimental)
  Interventions: Behavioral: Low FODMAP diet

INTERVENTIONS:
Behavioral: Low FODMAP diet — Low FODMAP diet instruction to irritable bowel syndrome patients.

SUMMARY:
Irritable bowel syndrome (IBS) is a common functional gastrointestinal disorder, affecting 15% of the population. IBS is characterized by recurrent abdominal pain/discomfort without identifiable organic lesions. The pathophysiology of IBS can be multi factors which included immune activation/inflammatory reactions, visceral hypersensitivity, gastrointestinal dysmotility, changes in gut microflora, brain-gut dysfunction and food intolerance. Many short-chain carbohydrates can induce abdominal symptoms, and these carbohydrates were called, Fermentable, Oligosaccharides, Disaccharides and Monosaccharides and Polyols (FODMAPs). Around 50- 86% of the IBS patients will have a clinically meaningful response to the low-FODMAP diet. To evaluate the efficacy of low FODMAP diet. Experimental design: Health control and patients meeting the ROME III criteria for IBS will be enrolled in this study. The basic profiles, patient characteristics, intestinal microbiota profiles and MRI images will be obtained before and after low FODMAP diet intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for the study if all of the following criteria are met:

1. Patients with irritable bowel syndrome as per Rome IV diagnostic criteria Symptom characteristics of IBS according to Rome III and IV criteria
2. Patients must provide witnessed written informed consent prior to any study procedures being performed
3. Patients aged between 20-65 years
4. Male or female patients

Exclusion Criteria:

* Exclusion criteria including:

  1. Unable to provide or understand written informed consent.
  2. Pregnancy.
  3. Receiving antibiotics or narcotics within 90 days prior to enrollment.
  4. Receiving new prebiotics, probiotics within 90 days prior to enrollment.
  5. Current infection.
  6. History of inflammatory bowel disease.
  7. Thyroid disease.
  8. Major psychiatric disorders, including clinical anxiety or depression and previous use of anxiolytics and antidepressants.
  9. Previous stroke, intracerebral hemorrhage, or central nervous system diseases.
  10. Malignancy.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
irritable bowel syndrome Severity Scale (IBS-SS) | Baseline, end of study approximately 6 to 8 weeks ]
  The primary endpoint is the variable used to assess the main objective, the efficacy of low FODMAP diet on gastrointestinal symptoms in IBS (focusing on the elimination phase) change from baseline after 6-8 weeks. The variables used will be the symptom scores of several symptom questionnaires. Ultimately, the efficacy of the diet is based on improvement of symptom scores. Improvement is defined as a 50-point drop on the Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS). In this questionnaire, each quesiton is scored from 0-100, with a maximum total score of 500. Patients reporting scores <50 are defined as non-IBS individuals, a score from 50-175 indicated mild disease, 175-300 moderate and >300 severe.